CLINICAL TRIAL: NCT06268717
Title: Understanding Gastrointestinal Alpha-Gal Syndrome: (GI Alpha-Gal Study)
Brief Title: GI Alpha-Gal Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Revivicor, Inc (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: 23-0316
Record Dates: First submitted 2024-02-12; First posted 2024-02-20 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Alpha-Gal Syndrome; Irritable Bowel Syndrome; Diarrhea; Abdominal Pain; Vomiting
Keywords: Alpha-Gal Syndrome; diarrhea; abdominal pain; vomiting
MeSH Terms: conditions — red meat allergy; Irritable Bowel Syndrome; Diarrhea; Abdominal Pain; Vomiting

STUDY DESIGN:
Intervention Model Description: Double-blind crossover. Each participant will be randomized to undergo two double-blind food challenges with at least a 10-day washout period between the challenges. One food challenge will contain pork meat containing alpha-gal sugar; one challenge will contain pork meat without alpha-gal sugar.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The principal investigator and clinical research coordinators will be blinded to the challenges during the course of the study. The metabolic kitchen and a delegated research staff member will be unblinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Food challenge with pork meat containing alpha-gal, then pork meat without alpha gal sugar (Active Comparator): Participants receive a food challenge, consuming pork meat that contains alpha-gal. After a >10-day washout period, participants undergo a food challenge with pork which does not contain alpha-gal.
  Interventions: Other: Ground pork containing alpha-gal; Other: Pork meat not containing alpha-gal
- Food challenge with pork meat without alpha gal sugar, then pork meat containing alpha-gal (Active Comparator): Participants receive a food challenge consuming pork meat that does not contain alpha-gal sugar. After a >10-day washout period, participants undergo a food challenge with pork which does contain alpha-gal.
  Interventions: Other: Ground pork containing alpha-gal; Other: Pork meat not containing alpha-gal

INTERVENTIONS:
Other: Ground pork containing alpha-gal — 150 grams of cooked, ground pork meat containing alpha-gal sugar eaten once
Other: Pork meat not containing alpha-gal — 150 grams of cooked, ground pork meat not containing alpha-gal sugar

SUMMARY:
This is a double-blind, crossover food challenge study using pork with and without α-gal in patients with a clinical diagnosis of gastrointestinal (GI)- α-gal allergy, and to investigate the pathophysiology underlying their symptoms.

DETAILED DESCRIPTION:
Each participant will be randomized to undergo two double-blind food challenges with at least a 10-day washout period between the challenges. One food challenge will contain pork meat with alpha gal sugar; one challenge will contain pork meat without the alpha gal sugar. During the challenges, participants will drink lactulose and C13 mannitol dissolved in water. The principal investigator and clinical research coordinators will be blinded to the challenges during the course of the study. The metabolic kitchen and a delegated research staff member will be unblinded.

On consenting patients, a transnasal upper endoscopy (TNE) will be performed on each challenge day, pre-challenge, at hour 0 and post-challenge, at hour 6. During the TNE, esophagus, stomach and small bowel samples will be collected. Gastrointestinal pathology samples will be evaluated for inflammatory cells and also biobanked for further messenger RNA (mRNA) sequencing studies.

Blood and urine will be collected during each challenge. Samples will be transported to a lab and analyzed for tryptase, basophil activation, and lactulose/ mannitol levels.

ELIGIBILITY:
Inclusion Criteria:

* The subject is at least 18 years of age.
* The subject has a history of gastrointestinal alpha-gal allergy defined by elevated test for α-gal allergy (α-gal IgE >0.1 U/L) due to complaints of either abdominal pain or discomfort, diarrhea, nausea with or without vomiting, or a combination of those complaints, within the last 5 years. The subjects must have experienced one or more of the four symptoms at least once monthly for at least two months. The subjects will fill out a symptom questionnaire of the presence of these four symptoms (abdominal pain or discomfort, diarrhea, nausea, vomiting), frequency and severity (mild, moderate, or severe) for the 3 months prior to diagnosis.
* The subject has experienced symptomatic improvement on a mammalian meat-free diet over at least a month's time, defined by saying "yes" to the following question: "On the alpha-gal avoidant diet, have you had adequate relief of gastrointestinal symptoms?"
* The subject has elevated α-gal IgE titer on screening for the trial if they do not have a positive titer within 6 months of enrollment.
* The subject is willing to not take nonsteroidal anti-inflammatory medications, leukotriene modifiers or steroids 14 days prior to challenge.
* The subject is willing to sign the informed consent form.

Exclusion Criteria:

* The subject has health conditions that would pose a significant threat in the face of anaphylaxis or treatment for anaphylaxis (e.g., cardiac disease, unstable angina pectoris, arrhythmias).
* The subject is allergic to mannitol.
* If female, the subject is pregnant.
* The subject has a history of chronic GI conditions, including inflammatory bowel disease, celiac disease, chronic pancreatitis with continued symptoms (experience moderate-severe abdominal pain, diarrhea, or nausea/vomiting that occur more frequently than once weekly)
* The subject has diarrhea (one or more loose stools that conform to the container), moderate to severe abdominal pain, or vomiting within 10 days prior to the challenge.
* The subject has a history of severe allergic reaction on mammalian meat ingestion (respiratory distress, chest pain or cardiopulmonary compromise)
* The subject is unwilling to receive intramuscular epinephrine.
* The subject is anticipated to use omalizumab within 6 months of enrollment.
* The subject is anticipated to use systemic steroids within 28 days of food challenge.
* The subject is anticipated to use leukotriene modifier within 14 days of food challenge.
* The subject is unable to not use nonsteroidal anti-inflammatory drugs for 14 days prior to challenge.

Additional Exclusion Criteria for Subjects Undergoing Transnasal Endoscopy and Biopsy

* Known conditions that are contraindications to transnasal endoscopy, or in the opinion of the investigator any condition that would interfere with the study objectives.
* History of head and neck malignancy or anatomical deformities of the nasopharynx
* Severe anxiety

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-10-17 (Actual); Primary Completion 2026-06-02 (Estimated); Study Completion 2026-06-02 (Estimated)

PRIMARY OUTCOMES:
Allergic reaction (food challenge positive) | 6 hours post ingestion
  Presence of allergic reaction within 6 hours of the challenge. Reported as dichotomous: food challenge positive (reaction) or food challenge negative (no reaction).
No allergic reaction (food challenge negative) | 6 hours post ingestion
  No allergic reaction within 6 hours of the challenge. Reported as dichotomous: food challenge positive (reaction) or food challenge negative (no reaction).
Lactulose excretion | 0- 6 hours post ingestion
  C13 mannitol quantification with high-performance liquid chromatography- C13 mannitol excreted in the urine in the six hours following ingestion will be measured as a marker of intestinal permeability.
C13 mannitol excretion | 0-6 hours post ingestion
  C13 mannitol quantification with high-performance liquid chromatography- C13 mannitol excreted in the urine in the six hours following ingestion will be measured as a marker of intestinal permeability.
Basophil activation threshold response at timepoint 0 | 0 hours (prior to ingestion)
  Basophil activation threshold responses - peripheral blood basophils will be isolated and stimulated with mammal-based extracts to create a dose-response curve for concentrations of antigen leading to CD63 activation
Basophil activation threshold response at 2 hours | 2 hours post ingestion
  Basophil activation threshold responses - peripheral blood basophils will be isolated and stimulated with mammal-based extracts to create a dose-response curve for concentrations of antigen leading to CD63 activation.
Basophil activation threshold response at 4 hours | 4 hours post ingestion
  Basophil activation threshold responses - peripheral blood basophils will be isolated and stimulated with mammal-based extracts to create a dose-response curve for concentrations of antigen leading to CD63 activation.
Basophil activation threshold response at 6 hours | 6 hours post ingestion
  Basophil activation threshold responses - peripheral blood basophils will be isolated and stimulated with mammal-based extracts to create a dose-response curve for concentrations of antigen leading to CD63 activation. Results pre- and post- pork challenge will be compared to assess for changes in basophil responses
Serum tryptase at timepoint 0 | 0 hours (prior to ingestion)
  Serum tryptase- serum tryptase levels will be quantified.
Serum tryptase at 2 hours | 2 hours post ingestion
  Serum tryptase- serum tryptase levels will be quantified.
Serum tryptase at 4 hours | 4 hours post ingestion
  Serum tryptase- serum tryptase levels will be quantified.
Serum tryptase at 6 hours | 6 hours post ingestion
  Serum tryptase- serum tryptase levels will be quantified.
Mast cell count on stomach biopsies (per high powered field (hpf)) | 6 hours post ingestion
  The number of mast cells will be counted at high-powered field on biopsy specimens of the stomach.
Mast cell count on small bowel biopsies (per high powered field (hpf)) | 6 hours post ingestion
  The number of mast cells will be counted at high-powered field on biopsy specimens of the small bowel.
Eosinophil cell count on stomach biopsies (per high powered field (hpf)) | 6 hours post ingestion
  The number of eosinophil cells will be counted at high-powered field on biopsy specimens of the stomach.
Eosinophil cell count on small bowel biopsies (per high powered field (hpf)) | 6 hours post ingestion
  The number of eosinophil cells will be counted at high-powered field on biopsy specimens of the small bowel.

SECONDARY OUTCOMES:
GI Symptom Rating Score (GSRS) | 24 hours post challenge
  The Gastrointestinal Symptom Rating Scale (GSRS) assesses gastrointestinal symptoms as experienced by participants in the 24-hours following a challenge. The scale covers 17 specific G1 symptoms, each rated on a 0-5 scale where 0 (no symptoms), 1 (very mild), 2 (mild), 3 (moderate), 4 (severe), 5 (very severe)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah McGill, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: beginning 9 and continuing for 36 months following publication
Access Criteria: Investigator has approved IRB, IEC, or REB and an executed data use/sharing agreement with UNC.